CLINICAL TRIAL: NCT06180785
Title: Performance Evaluation of the Biological Diagnosis of Heparin-induced Thrombocytopenia (HIT)
Brief Title: Performance Evaluation of the Biological Diagnosis of HIT
Acronym: HIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8665
Record Dates: First submitted 2022-09-06; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Heparin-induced Thrombocytopenia (HIT)
Keywords: Heparin-induced thrombocytopenia; HIT; heparin therapy; heparin treatments; molecular weight heparin; IgG antibodies; platelet factor 4 (PF4); heparin complex; thrombotic risk

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heparin-induced thrombocytopenia (HIT) is a severe complication of heparin therapy with a non-negligible incidence (estimated at 2.6% of unfractionated heparin treatments and 0.2% of low molecular weight heparin treatments). It is generally secondary to the appearance of IgG antibodies directed against the platelet factor 4 (PF4) - heparin complex. These antibodies, once bound to this complex, are likely to activate platelets: the thrombotic risk generated can be potentially fatal.

ELIGIBILITY:
Inclusion criteria :

* Adult patient (≥ 18 years of age)
* Hospitalized at HUS between 01/01/2009 and 31/12/2019
* Specimen sent to the HUS Hematology Laboratory for biological diagnosis of HIT between 01/01/2009 and 31/12/2019
* Data collected by the CRPV and analyzed by the HIT multidisciplinary group in order to reach a consensus decision on the presence or absence of HIT
* Patient does not object to the reuse of his medical data for scientific research purposes.

Exclusion criteria:

* Patient for whom no test has been performed at the HUS Hematology Laboratory
* Patient for whom no data has been collected by the CRPV
* Patient for whom the HIT group could not confirm or deny the presence of HIT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥ 18 years of age) hospitalized at HUS between 01/01/2009 and 31/12/2019
Sampling Method: Non-Probability Sample
Enrollment: 894 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of the biological diagnosis approach for heparin-induced thrombocytopenia (HIT) in the Hematology laboratory of the University Hospitals of Strasbourg | through study completion, an average of 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire d'Hématologie - CHU de Strasbourg - France, Strasbourg, France